CLINICAL TRIAL: NCT03347695
Title: A New Operation (Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure) for the Treatment of Long Standing Persistent Atrial Fibrillation (AF) During Mitral Valve Surgery
Brief Title: A New Operation for the Treatment for Long-standing Atrial Fibrillation
Acronym: ANOLAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, The director of the department of cardiovascular surgery, Fujian Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLW2017AF
Record Dates: First submitted 2017-11-11; First posted 2017-11-20 (Actual); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Disease
Keywords: atrial fibrillation; surgery
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A new operation (Experimental): Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure
  Interventions: Procedure: Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure(selected patients)
- A new operation (Selected pilot study) (Other): Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure
  Interventions: Procedure: Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure

INTERVENTIONS:
Procedure: Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure(selected patients) — Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure
  Arms: A new operation
Procedure: Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure — Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure
  Arms: A new operation (Selected pilot study)

SUMMARY:
Atrial fibrillation(AF) often occurs in patients with mitral valve disease. Both mitral replacement and mitral valve plasty are the effective methods to the mitral valve disease. How to cure atrial fibrillation is the key to full recovery. Radiofrequency ablation (RFA) in surgery is an effective treatment for those patients. But there are some recurrence rate after RFA, particularly in patients with enlarged left atrium. So the investigators design a new procedure(Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure) during mitral surgery and study the outcomes to evaluate this new operation.

DETAILED DESCRIPTION:
From September 2017, 20 selective patients, and then 120 consecutive patients with valvular atrial fibrillation were treated with our new operation. If the clinical results from the first 20 patients with restrict selection criteria are unsatisfied, that is, the restoration rate of the sinus rhythm was less than 50% at 1-year follow up, the study will be stopped. Otherwise, another single arm with 120 consecutive patients with valvular AF will be recruited for next phase.

Procedure details: All patients will have their left atrial geometric volume reduced, pulmonary vein island isolated and left appendage ligated or suture closed. After the superior vena cava was transected, two circular incisions were usually made in the left atrial wall between the pulmonary veins and the mitral annulus for circumferential atrial strip resection and pulmonary vein island isolation. The first circular incision was performed around the pulmonary veins. With this incision, pulmonary vein island was isolated and the left atrium was opened. The second one was performed in the interatrial groove and extended around the mitral annulus, leaving a 2 cm inferior wall margin from the annulus and the appendage in situ. With those two incisions, a circumferential strip of the left atrium was excised. Then the base of the left atrial appendage was ligated or excised and sutured. After the mitral manipulations, the center of the pulmonary vein island was longitudinally reef-imbricated with a 3-0 polypropylene continuous running suture to exclude toward the outside of the left atrial cavity. This plicated pulmonary vein island was directly anastomosed to the resected margin around the mitral annulus and the intraatrial septum instead of the interatrial groove. Finally, caval continuity was restored after aortic cross-clamp removal using a running 4-0 polypropylene suture.

Telephone contact was maintained with the patients after discharge.The use of antiarrhythmic medications will be allowed during the first 3 months(blanking period). Transthoracic 2-dimensional echocardiography and Holter monitoring will be obtained at baseline and at 3, 6, and 12 months after the initial operation. Whenever the participants have symptoms such as palpitation, dizziness, or shortness of breath, they could telephone the doctors.

The primary efficacy endpoint is freedom from AF at both 6 months and 12 months after surgery, assessed by 7-days continuous Holter monitoring. The primary safety are cardiopulmonary bypass time; and a composite of death, stroke, serious cardiac events (heart failure, myocardial infarction), cardiac re-hospitalizations, transient ischemic attack, pulmonary embolism, peripheral embolism, coronary artery injury, anatomical excessive bleeding, deep sternal wound infection/mediastinitis, damage to specialized conduction system requiring permanent pacemaker, and superior vena cava stenosis, within 30 days after the procedure or hospital discharge (whichever was later) The secondary efficacy endpoint are the left atrial linear dimensions and A wave reappearance measured by transthoracic echocardiography at 3 time points (before surgery, 6 and 12 months after surgery). The secondary safety endpoint are Major adverse cardiac events, which were defined as a non-weighted composite score of: death, stroke, worsening heart failure (+1 NYHA Class), hospitalization for heart failure, and mitral valve re-intervention within 12 months after surgery; and incidence of protocol-defined serious adverse events (especially thromboembolic and hemorrhagic events) within 12 months after surgery. Statistical analysis were performed with statistic package for social science( SPSS) 11.5 software. A value of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Phase I Inclusion Criteria

1. Able to sign Informed Consent and Release of Medical Information forms
2. Age ≥ 18 years and ≤ 60 years old
3. Clinical indications for only mitral valve surgery for the following:

   Organic mitral valve disease without other cardiac disorders (functional or structural).
4. Longstanding persistent AF is defined as continuous AF of greater than one year duration.

   Duration of AF must be documented by medical history and Presence of AF must be documented by a direct electrocardiographic assessment upon arrival in the clinic.
5. Able to use heart rhythm monitor
6. Anteroposterior diameter of left atrial between 45mm and 60mm
7. Without history of stroke. Exclusion Criteria

1. AF without indication for mitral valve surgery; or 2. Ischemic mitral regurgitation with evidence of concomitant structural mitral valve disease; or 3. Functional tricuspid regurgitation; or 4. AF is only or paroxysmal persistent; or 5. Evidence of active infection; or 6. Mental impairment or other conditions that may not allow patient to understand the nature, significance, and scope of study; or 7. Surgical management of hypertrophic obstructive cardiomyopathy; or 8. Previous catheter ablation for AF; or 9. Life expectancy of less than one year; or 10. Absolute contraindications for anticoagulation therapy; or 11. Enrollment in concomitant drug or device trials; or 12. Uncontrolled hypo- or hyperthyroidism; or 13. FEV1 < 30% of predicted value; or 14. Women who are pregnant as evidenced by positive pregnancy test; or 15. Women of childbearing age who do not agree to be on adequate birth control throughout the period of the trial; or 16. Diagnosed with infective endocarditis; or 17. Need emergency surgery. Phase II Inclusion Criteria

1. Able to sign Informed Consent and Release of Medical Information forms
2. Age ≥ 18 years
3. Clinical indications for mitral valve surgery for the following:

   Organic mitral valve disease; or Functional non-ischemic mitral regurgitation; or Ischemic mitral regurgitation with evidence of concomitant structural mitral valve disease.

   Note: May include need for surgical management of functional tricuspid regurgitation or patent foramen ovale. May also include concomitant CABG, aortic arch or aortic valve procedure. Surgical intervention may be performed via sternotomy or minimally invasive procedure.
4. Longstanding persistent AF is defined as continuous AF of greater than one year duration.

   Duration of AF must be documented by medical history and Presence of AF must be documented by a direct electrocardiographic assessment upon arrival in the clinic.
5. Able to use heart rhythm monitor

Exclusion Criteria

1. AF without indication for mitral valve surgery; or
2. AF is only or paroxysmal persistent; or
3. Evidence of active infection; or
4. Mental impairment or other conditions that may not allow patient to understand the nature, significance, and scope of study; or
5. Surgical management of hypertrophic obstructive cardiomyopathy; or
6. Previous catheter ablation for AF; or
7. Life expectancy of less than one year; or
8. Absolute contraindications for anticoagulation therapy; or
9. Enrollment in concomitant drug or device trials; or
10. Uncontrolled hypo- or hyperthyroidism; or
11. Women who are pregnant as evidenced by positive pregnancy test; or
12. Women of childbearing age who do not agree to be on adequate birth control throughout the period of the trial; or
13. Diagnosed with infective endocarditis; or
14. Need emergency surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liangwan Chen, M.D, Study Director — Union Hospital
Locations (1):
- Department of Cardiovascular Surgery,Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
plan to share study protocol, SAP and ICF with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the study ends.
Access Criteria: cardiovascular researchers
URL: http://www.fjxiehe.com

REFERENCES:
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Kim JH, Na CY, Lee SJ, Oh SS. Circumferential left atrium resection for treating a giant left atrium. J Card Surg. 2013 Mar;28(2):102-8. doi: 10.1111/jocs.12061. Epub 2013 Jan 29. PMID 23356418
- [Background] Shi J, Bai ZX, Zhang BG, Ren WJ, Guo YQ. A modified Cox maze IV procedure: a simpler technique for the surgical treatment of atrial fibrillation. Interact Cardiovasc Thorac Surg. 2016 Dec;23(6):856-860. doi: 10.1093/icvts/ivw256. Epub 2016 Aug 11. PMID 27521177
- [Background] Zheng S, Zhang H, Li Y, Han J, Jia Y, Meng X. Comparison of Left Atrial and Biatrial Maze Procedure in the Treatment of Atrial Fibrillation: A Meta-Analysis of Clinical Studies. Thorac Cardiovasc Surg. 2016 Dec;64(8):661-671. doi: 10.1055/s-0035-1554941. Epub 2015 Jul 28. PMID 26220695
- [Background] Kong MH, Lopes RD, Piccini JP, Hasselblad V, Bahnson TD, Al-Khatib SM. Surgical Maze procedure as a treatment for atrial fibrillation: a meta-analysis of randomized controlled trials. Cardiovasc Ther. 2010 Oct;28(5):311-26. doi: 10.1111/j.1755-5922.2010.00139.x. PMID 20370795
- [Background] Baek MJ, Na CY, Oh SS, Lee CH, Kim JH, Seo HJ, Park SW, Kim WS. Surgical treatment of chronic atrial fibrillation combined with rheumatic mitral valve disease: Effects of the cryo-maze procedure and predictors for late recurrence. Eur J Cardiothorac Surg. 2006 Nov;30(5):728-36. doi: 10.1016/j.ejcts.2006.08.016. Epub 2006 Sep 26. PMID 17008109
- [Background] Kumar P, Athanasiou T, De L Stanbridge R. Treatment of long-duration atrial fibrillation by modified maze procedure. J R Soc Med. 2002 Nov;95(11):552-3. doi: 10.1258/jrsm.95.11.552. No abstract available. PMID 12411621
- [Derived] Chen L, Li Q, Chen J, Qiu Z, Xiao J, Tang M, Wu Q, Shen Y, Dai X, Fang G, Lu H. A new procedure for elimination of atrial fibrillation associated with mitral valve disease: a proof-of-concept study. Int J Surg. 2023 Oct 1;109(10):2914-2925. doi: 10.1097/JS9.0000000000000566. PMID 37352525

RESULTS

PARTICIPANT FLOW:
Groups:
- A New Operation (Selected Pilot Study): Two circular incisions were performed in the left atrial wall between the pulmonary veins and the mitral annulus. with those two incisions, circumferential resection of a strip for the left atrial was obtained. The middle of pulmonary vein island was longitudinal plicated and the left appendage was ligated. Finally,the plicated pulmonary island was directly anastomosed to the lest side free wall, inferior wall, roof, the posterior walls of both superior and inferior vein cavae, and intra-atrial septum.
  Left atrial geometric volume reduction, pulmonary veins island isolation and left appendage ligation (Selected): Two circular incisions were performed in the left atrial wall between the pulmonary veins and the mitral annulus. with those two incisions, circumferential resection of a strip for the left atrial was obtained. The middle of pulmonary vein island was longitudinal plicated and the left appendage was ligated. Finally,the plicated pulmonary island was directly anastomosed to the lest side free wall, inferior wall, roof, the posterior walls of both superior and inferior vein cavae, and intra-atrial septum.
- A New Operation: Two circular incisions were performed in the left atrial wall between the pulmonary veins and the mitral annulus. with those two incisions, circumferential resection of a strip for the left atrial was obtained. The middle of pulmonary vein island was longitudinal plicated and the left appendage was ligated. Finally,the plicated pulmonary island was directly anastomosed to the lest side free wall, inferior wall, roof, the posterior walls of both superior and inferior vein cavae, and intra-atrial septum.
  Left atrial geometric volume reduction, pulmonary veins island isolation and left appendage ligation: Two circular incisions were performed in the left atrial wall between the pulmonary veins and the mitral annulus. with those two incisions, circumferential resection of a strip for the left atrial was obtained. The middle of pulmonary vein island was longitudinal plicated and the left appendage was ligated. Finally,the plicated pulmonary island was directly anastomosed to the lest side free wall, inferior wall, roof, the posterior walls of both superior and inferior vein cavae, and intra-atrial septum.
Period: Overall Study
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Started | 20 | 120
Completed | 20 | 115
Not Completed | 0 | 5
Not completed — Death | 0 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation | Total
Number analyzed (Participants) | 20 | 120 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 113 | 133
  >=65 years | 0 | 7 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (9.6) | 52.3 (8.0) | 51.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 74 | 87
  Male | 7 | 46 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 120 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 20 | 120 | 140
Hypertension [Count of Participants; unit: Participants] | 1 | 13 | 14
Prior stroke [Count of Participants; unit: Participants] | 0 | 12 | 12
Diabetes [Count of Participants; unit: Participants] | 1 | 5 | 6
Smoking History [Count of Participants; unit: Participants] | 2 | 25 | 27
NYHA Class III or Class IV [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification is used to classify patients' heart failure according to the severity of their symptoms. Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases. Class III and Class IV indicate worse heart function than Class I or Class II, and increase the risk of death for cardiac surgery.
  Participants | 20 | 112 | 132
Long-standing persistent AF [Count of Participants; unit: Participants] | 20 | 120 | 140
Atrial fibrillation duration [Mean (Standard Deviation); unit: months] | 19.4 (6.5) | 23.6 (9.7) | 23.0 (9.4)
EuroScore [Mean (Standard Deviation); unit: units on a scale] — European system for cardiac operative risk evaluation (EuroSCORE) is a scoring system for the prediction of early mortality in cardiac surgical patients. It is the sum of several scored patients-related fators, such as, age, sex, comorbidities and operation information, and so on. Usually, the low risk group is defined as EuroSCORE 1-2 with 0.8% deaths risk, 3% for medium risk group (EuroSCORE 3-5), 11.2% for high risk group (EuroSCORE 6 plus). The range of EuroSCORE in this study is from 0 to 22.
  units on a scale | 1.8 (1.6) | 1.8 (1.4) | 1.8 (1.4)
Preoperative amiodarone intake [Count of Participants; unit: Participants] | 1 | 3 | 4
Preoperative Digoxin intake [Count of Participants; unit: Participants] | 11 | 69 | 80
Preoperative beta-blocker intake [Count of Participants; unit: Participants] | 5 | 23 | 28
Preoperative NT-proBNP level [Mean (Standard Deviation); unit: pg/ml] | 1555.3 (1233.2) | 1482.3 (1321.8) | 1493.0 (1305.0)
Preoperative creatine level [Mean (Standard Deviation); unit: μmol/l] | 77.5 (16.3) | 79.4 (44.9) | 79.1 (42.0)
left ventricular diastolic diameter [Mean (Standard Deviation); unit: milimeters] | 48.7 (7.0) | 49.7 (7.5) | 49.6 (7.4)
left ventricular systolic diameter [Mean (Standard Deviation); unit: milimeters] | 34.0 (5.7) | 33.6 (5.7) | 33.7 (5.7)
left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 57.1 (8.1) | 60.5 (8.7) | 60.0 (8.7)
left atrial anteroposterior diameter [Mean (Standard Deviation); unit: milimeters] | 55.0 (3.3) | 54.8 (9.3) | 54.9 (8.7)
left atrial transversal diameter [Mean (Standard Deviation); unit: milimeters] | 59.4 (6.3) | 59.6 (13.1) | 59.6 (12.4)
left atrial superoinferior diameter [Mean (Standard Deviation); unit: milimeters] | 68.9 (6.3) | 72.0 (15.4) | 71.5 (14.5)
Mitral Lesion [Count of Participants; unit: Participants] | 20 | 120 | 140
Aortic Lesion [Count of Participants; unit: Participants] | 0 | 58 | 58
Tricuspid Lesion [Count of Participants; unit: Participants] | 0 | 85 | 85
Coronary Heart Disease [Count of Participants; unit: Participants] | 0 | 3 | 3
mitral valve procedure [Count of Participants; unit: Participants]
  mitral valve replacement | 20 | 109 | 129
  mitral valve repair | 0 | 11 | 11
aortic valve replacement [Count of Participants; unit: Participants] | 0 | 35 | 35
Tricuspid valve repair [Count of Participants; unit: Participants] | 0 | 38 | 38
Concomitant CABG [Count of Participants; unit: Participants] | 0 | 3 | 3
Total surgery time [Mean (Standard Deviation); unit: minutes] | 221.6 (33.9) | 230.7 (48.4) | 229.4 (46.6)
aortic cross-clamp duration [Mean (Standard Deviation); unit: minutes] | 44.4 (17.8) | 52.5 (23.5) | 51.4 (22.9)
Total cardiopulmonary bypass time [Mean (Standard Deviation); unit: minutes] | 95.5 (19.0) | 106.8 (33.4) | 105.2 (31.9)

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants Free From AF
Description: Freedom from AF in patients with longstanding persistent AF undergoing MVS at 6 months and 12 months. AF will be measured by 7 days continuous Holter monitoring at 6 months and 12 months post-surgery; and freedom of AF will be defined by absence of AF lasting > 30 seconds at 12 months
Time Frame: 3, 6, and 12 months after the operation
Population: Twenty patients were enrolled in pilot study and 120 patients were enrolled in latter prospective study.
Measure: Count of Participants; unit: Participants
Groups:
- A New Operation (Selected Pilot Study): Left Atrial Geometric Volume Reduction, Pulmonary Vein Island Isolation and Left Appendage Base Closure(selected patients)
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 120
Participants
  at discharge | 20 | 96
  3 months after the operation | 20 | 97
  6 months after the operation | 20 | 97
  12 months after the operation | 20 | 98

2. Primary Outcome: Intraoperative Cardiopulmonary Bypass Duration
Description: Cardiopulmonary bypass (CPB) technology is used in most cardiovascular surgeries. These surgeries utilize CPB, which has been associated with some adverse effects. This is most likely due to exposure of blood to abnormal surfaces and conditions leading to systemic inflammatory responses. Prolonged CPB duration is associated with worse clinical outcomes.
Time Frame: 1 hour after operation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 120
minutes | 44.4 (17.8) | 52.5 (23.5)

3. Primary Outcome: The Adverse Events Within 30 Days After Surgery
Description: The adverse events within 30 days after surgery, including: death, stroke, serious cardiac events (heart failure, myocardial infarction), cardiac re-hospitalizations, transient ischemic attack, pulmonary embolism, peripheral embolism, coronary artery injury, anatomical excessive bleeding, deep sternal wound infection/mediastinitis, damage to specialized conduction system requiring permanent pacemaker, and superior vena cava stenosis.
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 120
Participants
  death | 0 | 2
  stroke | 0 | 1
  serious cardiac events (heart failure, myocardial infarction) | 0 | 1
  deep sternal wound infection/mediastinitis | 0 | 1
  transient ischemic attack, pulmonary embolism, peripheral embolism | 0 | 0
  coronary artery injury | 0 | 0
  anatomical excessive bleeding | 0 | 0
  damage to specialized conduction system requiring permanent pacemaker | 0 | 0

4. Secondary Outcome: Change in Left Atrial Anteroposterior Diameter
Description: echocardiographic change in left atrial anteroposterior diameter
Time Frame: 6 months and 12 months post-surgery
Population: Twenty patients were enrolled in pilot study and 120 patients were enrolled in latter prospective study. Two of 120 patients died in 30d after surgery，leaving 118 patients to be included in this cohort.
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 118
milimeters
  6 months post-surgery: number analyzed (Participants) | 20 | 116
  6 months post-surgery | 37.0 (3.0) | 39.6 (6.7)
  12 months post-surgery: number analyzed (Participants) | 20 | 115
  12 months post-surgery | 36.8 (3.1) | 39.2 (6.7)

5. Secondary Outcome: Change in Left Atrial Transversal Diameter
Description: echocardiographic change in left atrial transversal diameter
Time Frame: 6 months and 12 months post-surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 118
milimeters
  6 months post-surgery: number analyzed (Participants) | 20 | 116
  6 months post-surgery | 40.5 (4.6) | 42.1 (7.6)
  12 months post-surgery: number analyzed (Participants) | 20 | 115
  12 months post-surgery | 40.3 (4.7) | 42.5 (7.7)

6. Secondary Outcome: Change in Left Atrial Superoinferior Diameter
Description: echocardiographic change in left atrial superoinferior diameter
Time Frame: 6 months and 12 months post-surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 118
milimeters
  6 months post-surgery: number analyzed (Participants) | 20 | 116
  6 months post-surgery | 50.3 (3.6) | 54.7 (8.2)
  12 months post-surgery: number analyzed (Participants) | 20 | 115
  12 months post-surgery | 50.3 (3.8) | 55.7 (8.4)

7. Secondary Outcome: The Number of Participants Who Will be Detected the Peak Late Trans-mitral Flow Velocity (A Wave) Reappearance
Description: The peak late trans-mitral flow velocity (A wave) reappearance means recover of efficient left atrial contraction which indicates lower rate of thrombosis. Usually these is no A wave for AF patients. The peak late trans-mitral flow velocity 6 months and 12 months post-surgery, which will be measured by transthoracic echocardiography.
Time Frame: 6 months and 12 months post-surgery
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 118
Participants
  peak late trans-mitral flow velocity (A) reappearance rate 6 months post-surgery: number analyzed (Participants) | 20 | 97
  peak late trans-mitral flow velocity (A) reappearance rate 6 months post-surgery | 18 | 80
  peak late trans-mitral flow velocity (A) reappearance rate 12 months post-surgery: number analyzed (Participants) | 20 | 98
  peak late trans-mitral flow velocity (A) reappearance rate 12 months post-surgery | 18 | 84

8. Secondary Outcome: MACEs Within 12 Months After Surgery
Description: MACEs within 12 months after surgery: defined as a non-weighted composite score of: death, stroke, worsening heart failure (+1 NYHA Class), CHF hospitalization, and mitral valve [MV] re-intervention.
Time Frame: Within 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
Number analyzed (Participants) | 20 | 118
Participants
  death: number analyzed (Participants) | 20 | 117
  death | 0 | 2
  stroke: number analyzed (Participants) | 20 | 117
  stroke | 0 | 3
  worsening heart failure (+1 NYHA Class): number analyzed (Participants) | 20 | 117
  worsening heart failure (+1 NYHA Class) | 0 | 1
  mitral valve [MV] re-intervention: number analyzed (Participants) | 20 | 117
  mitral valve [MV] re-intervention | 0 | 1
  Pacemaker implantation: number analyzed (Participants) | 20 | 117
  Pacemaker implantation | 0 | 1

ADVERSE EVENTS:
Time Frame: Within 12 Months After Surgery
Description: in-hospital mortality rate, stroke or transient ischemic attack(TIA), heart failure, permanent pacemaker implantation, renal failure, pneumonia, sepsis, respiratory failure, and multiple organ dysfunction syndrome, which are defined by protocol within 12 months after surgery.
Arm/Group | A New Operation (Selected Pilot Study) | A New Operation
All-Cause Mortality (participants affected / at risk) | 0/20 | 4/120
Serious Adverse Events (participants affected / at risk) | 1/20 | 24/120
Other Adverse Events (participants affected / at risk) | 0/20 | 2/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A New Operation (Selected Pilot Study) (N=20) | A New Operation (N=120)
30-day (in-hospital) mortality (General disorders) | 0 (0) | 2 (2)
stroke or transient ischemic attack(TIA) (Nervous system disorders) | 0 (0) | 4 (4) — All stroke or transient ischemic attack(TIA) events within 12 months after surgery
heart failure (Cardiac disorders) | 0 (0) | 1 (1) — All heart failure events within 12 months after surgery
permanent pacemaker implantation (Cardiac disorders) | 0 (0) | 1 (1) — All permanent pacemaker implantation events within 12 months after surgery
renal failure (Renal and urinary disorders) | 0 (0) | 4 (4) — All renal failure events within 12 months after surgery
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) — All pneumonia within 12 months after surgery
sepsis (Infections and infestations) | 0 (0) | 1 (1) — All sepsis events within 12 months after surgery
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — All respiratory failure events within 12 months after surgery
multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2) — All multiple organ dysfunction syndrome events within 12 months after surgery
Reoperation (Surgical and medical procedures) | 0 (0) | 1 (1) — All reoperation events within 12 months after surgery
deep sternal infection (Infections and infestations) | 0 (0) | 1 (1) — All deep sternal infection events within 12 months after surgery
infective endocarditis (Cardiac disorders) | 0 (0) | 1 (1) — All infective endocarditis events within 12 months after surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A New Operation (Selected Pilot Study) (N=20) | A New Operation (N=120)
superficial wound infection (Infections and infestations) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03347695/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form for phase1 (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03347695/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form for phase2 (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03347695/ICF_002.pdf